CLINICAL TRIAL: NCT06956027
Title: Ultrasound Features of Dupuytren's Disease: Echogenicity, Skin Involvement and Microvascularisation
Brief Title: Ultrasound Features of Dupuytren's Disease
Acronym: Micro in DD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S70180
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Dupuytren disease (Other): Population of Dupuytren's Disease patients who fulfill study criteria
  Interventions: Diagnostic Test: Ultrasound assesment; Procedure: ROM measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound assesment — Ultrasound image taken using MV-flow technique for measuring the distance skin-lesion and echogenicity measurement
Procedure: ROM measurement — Range Of Motion measurement of affected finger(s) where the ultrasound image will be taken from.

SUMMARY:
Dupuytren's disease (DD) is a benign and progressive condition that affects the palmar aponeurosis with a very high global incidence. It can result in significant loss of hand function or can inhibit an individual's daily activities or work. Current diagnostics rely on Range Of Motion (ROM) measurements and clinical expertise, where the decision for treatment is primarily based on patient preferences with little scientific research supporting different options in different cases.

With technological advancements new options arise to the possible diagnostic tools we can use for evidence based medicine and shared decision making. One option comes to light for DD because of its cheap, non -invasive and no radiation load, namely ultrasound (US). The use of US for DD is not standard care, due to the lack of research surrounding this tool. This study will provide some insight into the use of US for DD and will primarily try to evaluate different parameters measurable with US that can be used as potential prognostic biomarkers.

DETAILED DESCRIPTION:
Dupuytren's disease (DD) is a benign and progressive condition that affects the palmar aponeurosis with a very high global incidence. It can result in significant loss of hand function or can inhibit an individual's daily activities or work. The diagnostic tool that is currently used the most is the clinical evaluation of a hand surgeon, and also the use of a goniometer which measures the total Range of Motion (ROM) a patient still has in his finger, where the decision for treatment is primarily based on patient preferences with little scientific research supporting different options in different cases. Due to a lack of patient satisfaction and high recurrence rates among those who underwent surgery there is a clear need for more knowledge surrounding DD to better understand this disease. This will lead to new possibilities in the field of research and the potential for new treatments.

With technological advancements new options arise to the possible diagnostic tools we can use for evidence based medicine and shared decision making. One option comes to light for DD because of its cheap, non -invasive and no radiation load, namely ultrasound (US). The use of US for DD is not standard care, due to the lack of research surrounding this tool. This study will provide some insight into the use of US for DD and will primarily try to evaluate different parameters measurable with US that can be used as potential prognostic biomarkers. Three different characteristics will be measured: echogenicity, skin involvement, the presence of microvascular structures. In summary, the mentioned parameters could possibly prove to be useful in the assessment of DD patients and could make US a standard in determining disease progression and could make the consideration between different treatment options more evidence based.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Clinical diagnosis of DD and a Tubiana staging not exceeding stage II, TPED does not exceed 90°; this is chosen because to great of a contracture will pose problems with taking the US measurement.
3. In the clinical assessment the subject has rather soft DD nodules, more firm nodules are more fibrotic and are less likely to contain blood vessels. This will be confirmed by a hand surgeon at the screening phase.
4. Participant has self reported rapid progression. In the anamnesis the subject reports one of the following: The DD lesion has changed in degree of contracture/nodule size recently; the patient is worried about the function of the involved fingers/hand due to recent progression; the patient is new to DD or has just started experiencing greater discomfort due to a previous existing nodule.
5. Participant agrees to not undergo any form of surgical treatment for DD during the duration of their participation, being 6 months.
6. Participant agrees to return to the clinic after 6 months voluntarily for follow-up measurements.

Exclusion Criteria:

1. Participant has any other disorder or pathology of the hand/fingers that could affect the quality of US measurements. This list is exhaustive: trigger finger, fracture, hematoma, tenosynovitis, tendon ruptures, scleroderma, fibromatosis, inflammatory conditions, rheumatoid arthritis, osteoarthritis.
2. Participant has received prior treatment for Dupuytren's disease (needle fasciotomy, (micro)fasciectomy) in the hand under investigation.
3. Participant's affected finger exceeds a TPED over 90° (= Tubiana stage III) (this will affect the value of any US images taken)
4. Participant undergoes treatment for DD during the course of their participation in this study: exhaustive list: fasciectomy/fasciotomy/stretching braces/collagenase injections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Echogenicity | At screening and at 6 month follow-up visit
  A biomarker measured with an ultrasound device that shows high myofibroblast presence (=hypoechogenic) or high collagen in the extracellular matrix (mean gray value).
Distance from the Duputren's Disease lesion to the skin | At screening and at 6 month follow-up visit
  This measurement shows skin involvement in the disease which will influence how it evolves (in millimeters).
Microvascularisation | At screening and at 6 month follow-up visit
  Determine the presence of microvascularisation inside the DD nodule. The presence of this vascularisation could be indicative of faster progression. (Answered with Yes or No)
Disease progression determined by TPED increase after 6 months | At screening and at 6 month follow-up visit
  The Total Passive Extension Deficit (PED) will be measured using a digital goniometer (in degrees). Disease progression when increase is ≥ 5°
Disease progression determined by URAM increase after 6 months | At screening and at 6 month follow-up visit
  The URAM questionnaire is used to determine progression for subject's own experience with the disease. Disease progression if URAM questionnaire score increases with 1 or more points (answered with Yes or No)

SECONDARY OUTCOMES:
Diathesis score | At screening and at 6 month follow-up visit
  This score goes from 0 till 9. To investigate if a high score (≥ 4) correlates with faster disease progression.
Incidence of the presence of microvascularisation | At screening and at 6 month follow-up visit
  The amount of participants with microvascularisation (given in %)

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No